CLINICAL TRIAL: NCT02128009
Title: Study on the Molecular Mechanism in Postmenopausal Osteoporosis With Kidney Yin Deficiency Syndrome Based on miRNA Mediated Gene Translation Regulation Function by Targeting CLCF1
Brief Title: Study on the microRNA Expression Level in Postmenopausal Osteoporosis
Acronym: microRNA
Status: Completed | Type: Observational
Sponsor: Fujian Academy of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-2-73
Record Dates: First submitted 2014-03-14; First posted 2014-05-01 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- osteoporosis,non-osteoporosis
  Interventions: Other: osteoporosis

INTERVENTIONS:
Other: osteoporosis

SUMMARY:
The miRNA plays an important regulation role in gene expression, and also closely related to bone metabolism. Previous research found that postmenopausal osteoporosis with kidney Yin deficiency syndrome (POP) is associated with CLCF1 gene. This project proposed by bioinformatics prediction CLCF1 targeted regulation of miRNAs, and use the 3 'UTR dual luciferase report system for target validation, aimed at the miRNA levels to explore postmenopausal osteoporosis molecular mechanism with kidney Yin deficiency syndrome.

ELIGIBILITY:
Inclusion Criteria:

* The Participants who volunteer to be test subjects, and can accept experimental drugs, and promise to finish the course should sign the informed consent.
* Female ages 45 to 75 had gone through natural menopause before two years
* In accordance with the western medicine diagnostic criteria of osteoporosis and belong to kidney Yin deficiency syndrome differentiation of traditional Chinese medicine certificate;
* In accordance with the western medicine diagnostic criteria;
* In accordance with TCM diagnostic methods; .If any of the above answers are no, The subjects couldn't in the study.

Exclusion Criteria:

* Do not accord with standard of the western medicine diagnosis and TCM diagnostic methods
* Age: <44 and > 76 years old;
* With hyperparathyroidism, osteomalacia, rheumatoid arthritis, multiple myeloma and other serious complications such as secondary osteoporosis; Late or deformity, disability, loss of labor;
* With cardiovascular, cerebrovascular, liver, kidney and hematopoietic system and other serious primary diseases;
* Psychosis or alzheimer's patients;
* Nearly three months, the use of hormone replacement therapy (HRT) and taking calcitonin, nearly six months has used double phosphonic acid salt for 15 days, etc.;
* This medicine allergic constitution or composition of known to have allergies;
* In a critical condition, It's difficult to make exact evaluators to efficacy and safety of the new drugs;

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatient clinic
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
microRNA expression lever in the Peripheral Blood | one year

CONTACTS AND LOCATIONS:
Overall Officials: FJ ITCM, provincial, Principal Investigator — Fujian Institute of Trational Chiness Medicine
Locations (1):
- Fujian Institute of Trational Chiness Medicine, Fuzhou, Fujian, China

REFERENCES:
- [Background] McClung MR, Grauer A, Boonen S, Bolognese MA, Brown JP, Diez-Perez A, Langdahl BL, Reginster JY, Zanchetta JR, Wasserman SM, Katz L, Maddox J, Yang YC, Libanati C, Bone HG. Romosozumab in postmenopausal women with low bone mineral density. N Engl J Med. 2014 Jan 30;370(5):412-20. doi: 10.1056/NEJMoa1305224. Epub 2014 Jan 1. PMID 24382002